CLINICAL TRIAL: NCT03681925
Title: The Effects of Nutrition Literacy Assessment on Patient-Centered Nutrition Education Provided by Dietitians
Brief Title: Measuring Nutrition Literacy in Clinical Practice: Evaluating Effects Upon Providers and Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: STUDY00142818
Record Dates: First submitted 2018-09-14; First posted 2018-09-24 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: Patient-centered care; Dietitian; Nutrition literacy
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: 6 dietitians will be randomized in a 2:1 intervention:control fashion. Each dietitian will recruit 19 patient participants, for 114 total patient participants.
Who Masked: Participant
Masking Description: Patient participants will be unaware of which arm their dietitian has been randomized to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Dietitians randomized to the intervention arm will have access to their participating patients' Nutrition Literacy Assessment Instrument (NLit) scores, and base their intervention on these results.
  Interventions: Diagnostic Test: Nutrition Literacy Assessment Instrument (NLit)
- Control (No Intervention): Dietitians randomized to the control arm will not have access to their participating patients' Nutrition Literacy Assessment Instrument (NLit) scores, and will provide the standard-of-care intervention for their patients.

INTERVENTIONS:
Diagnostic Test: Nutrition Literacy Assessment Instrument (NLit) — The NLit is a 64-question survey broken into 6 subscales. each subscale examines a different aspect of nutrition literacy (Nutrition and Health, Energy Sources in Food, Household Food Measurement, Food Label and Numeracy, Food Groups, and Consumer Skills). Global and subscale NLit scores will be generated for each participating patient.
  Arms: Intervention

SUMMARY:
This study evaluates the effects of assessing patient nutrition literacy prior to an initial session with an outpatient dietitian on the patient-centeredness of the session. We will randomize 6 dietitians, 4 of whom will have access to their participating patients' nutrition literacy scores. These dietitians will use this information to better inform their interventions, and hopefully improve their patients' nutrition literacy as a result.

DETAILED DESCRIPTION:
Nutrition Literacy Assessment Tool (NLit): a validated, 64-question survey that assesses nutrition literacy across 6 subscales:

* Nutrition and Health
* Energy Sources in Food
* Household Food Measurement
* Food Label and Numeracy
* Food Groups
* Consumer Skills

Dietitians who work within 6 different outpatient clinics (1 dietitian per clinic) will be recruited to the study; each dietitian will recruit 19 patients from their clinic. All patient participants will take the NLit survey prior to an initial visit with their dietitian. Dietitians randomized to the intervention arm (n=4) will have access to their participating patients' NLit results, and tailor their intervention to the patient's nutrition literacy weaknesses. Dietitians randomized to the control group (n=2) will not have access to their participating patients' NLit scores, and will provide the same standard-of-care intervention usually provided.

All participating patients will then re-take the NLit a month after their initial session with their dietitian, and we will examine the results to see if a) nutrition literacy improved within groups, and b) if the patients of the intervention dietitians showed more improvement in nutrition literacy than their counterparts being treated by the control dietitians.

We will also collect dietary pattern information from participating patients before their initial session with their dietitian, and again one month after their initial session with their dietitian. We will examine the results to see if a) dietary patterns improve with increased nutrition literacy, and b) if the dietary patterns of patients in the intervention group improve more than patients in the control group.

Finally, we will collect survey information from patients pertaining to the perceived patient-centeredness of the session with their dietitian. We will also collect audio recordings of the sessions between patients and dietitians, which will be analyzed for patient-centeredness. We will also analyze readability and clearness of printed materials used by dietitians during their interventions with patients.

ELIGIBILITY:
Inclusion Criteria:

* subjects must be at least 18 years old
* subjects must be able to read English
* subjects must be scheduled with a participating dietitian

Exclusion Criteria:

* subjects with cognitive disabilities or overt mental illnesses
* subjects with vision issues severe enough to disrupt reading of the NLit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Change in Nutrition Literacy Assessment Instrument (NLit) score from baseline to post-session. | Nutrition literacy will be measured prior to the patients' initial session with a dietitian, then again one month after the session.
  Nutrition literacy will be assessed with the Nutrition Literacy Assessment Instrument (NLit)

SECONDARY OUTCOMES:
Change in BRFSS 2011 Fruit and Vegetable Module scores from baseline to one month post-session. | BRFSS 2011 Fruit and Vegetable Module scores will be measured prior to the patients' initial session with a dietitian, then again one month after the session.
  Dietary patterns will be assessed using the BRFSS 2011 Fruit and Vegetable Module.
Change in Rapid Eating Assessment for Patients (REAP) score from baseline to one month post-session | BRFSS 2011 Fruit and Vegetable Module scores will be measured prior to the patients' initial session with a dietitian, then again one month after the session.
  Dietary patterns will be assessed using the Rapid Eating Assessment for Patients (REAP)
Patient view of patient-centeredness of the session with a dietitian | Patients will complete the survey up to two months after they complete their session with a dietitian.
  Patient view of patient-centeredness of the session will be assessed using a modified version of the Consumer Assessment of Healthcare Providers and Systems-Clinician and Group Survey (CAHPS), v.3.0
Patient-centeredness of the session between patient and dietitian | One month post-session
  Patient-centeredness of the session between patient and dietitian will be assessed using the Teach back Loop Score, a validated tool used to examine the use of teach back, an essential part of patient-centered care.
Readability of printed materials used by dietitians during interventions | One month prior to first patient session with a dietitian
  Reading level of all printed materials will be assessed using the Flesch-Kincaid Readability score.
Clearness of printed materials used by dietitians during interventions | One month prior to first patient session with a dietitian
  Clearness of printed materials will be assessed using the Center for Disease Control Clear Communications Index

CONTACTS AND LOCATIONS:
Overall Officials: Heather D Gibbs, PhD, Principal Investigator — University of Kansas Medical Center
Locations (5):
- United States (5):
  - The University of Kansas Health System Family Medicine and Internal Medicine Clinics, Kansas City, Kansas
  - University of Kansas Medical Center Student Health Services, Kansas City, Kansas
  - University of Kansas Medical Center, Center for Physical Activity and Weight Management, Kansas City, Kansas
  - University of Kansas Medical Center Bariatric and Weight Loss Surgery Clinic, Overland Park, Kansas
  - Encompass Medical Group, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gibbs HD, Ellerbeck EF, Gajewski B, Zhang C, Sullivan DK. The Nutrition Literacy Assessment Instrument is a Valid and Reliable Measure of Nutrition Literacy in Adults with Chronic Disease. J Nutr Educ Behav. 2018 Mar;50(3):247-257.e1. doi: 10.1016/j.jneb.2017.10.008. Epub 2017 Dec 12. PMID 29246567